CLINICAL TRIAL: NCT06136299
Title: Effect of Neuromuscular Training on Physical Performance and Injury Rate in Elite Female Youth Soccer Players
Brief Title: Neuromuscular Training in Female Youth Soccer
Acronym: NMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Shari Liberman, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00036803
Record Dates: First submitted 2023-11-01; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Injury;Sports
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Intervention Model Description: There are two groups for this study. The control group performs their standard warm-up during soccer practice sessions and the experimental group performs neuromuscular training (NMT) in the form of the FIFA 11+ Kids program as their warm up.
Who Masked: Outcomes Assessor
Masking Description: All staff members measuring performance at the pre- and post-intervention testing sessions were unaware of which group the subject was randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Standard warm-up (No Intervention): This group performed a standard warm-up protocol during their soccer practice sessions.
- Intervention - NMT (Experimental): This group performed a specific Neuromuscular Training (NMT) warm-up program known as FIFA 11+ Kids during their soccer practice sessions
  Interventions: Other: Neuromuscular Training

INTERVENTIONS:
Other: Neuromuscular Training — This intervention uses the FIFA 11+ Kids program as a warm-up during soccer practice sessions.
  Arms: Intervention - NMT

SUMMARY:
The goal of this clinical trial is to analyze the effectiveness of an NMT-based, injury prevention training program ('FIFA 11+ for Kids') in pre-adolescent (Ages 8 to 11) elite female soccer players by measuring neuromuscular control and motor coordination through pre-intervention and post-intervention testing. As well as monitoring the incidence of injury throughout a soccer season.

DETAILED DESCRIPTION:
This study will recruit females aged between 8-11 from several teams within a large, competitive elite soccer club. Whole teams will be assigned to either the intervention group or an age-matched control group. Participants will be informed which group they will be placed in prior to participation in the research study. As directed by their respective coaches, the intervention group will receive neuromuscular training (NMT) through an already established, validated protocol (FIFA 11+ Kids); whilst the control group will perform their standard warm-up during soccer practice sessions. The program will last for the duration of the spring soccer season (January - May 2023; 5 months). All study participants will be required to attend two evaluation sessions (pre-intervention and post-intervention) in order to measure performance in speed, agility, hop testing, dynamic balance and strength.

ELIGIBILITY:
Inclusion Criteria:

* Elite female soccer players aged 8-11.
* Member of an elite youth soccer club.

Exclusion Criteria:

* Female not aged 8-11 years old.
* Not a member of a youth soccer club.
* Unable to attend the pre-intervention or post-intervention evaluation, for reasons other than injury.
* Unable to attend 80% or more of scheduled training sessions.
* If a participant discontinues playing soccer they will be excluded.
* Declines to participate in study.

Ages: 8 Years to 11 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Dynamic balance assessment | Dynamic balance will be measured at two separate timepoints: pre-intervention (baseline) and post-intervention (within 5-months after baseline measures).
  The Y-balance test is a standardized protocol consisting of lower extremity reach in the anterior, posteromedial and posterolateral directions.
Strength assessment | Strength will be measured at two separate timepoints: pre-intervention (baseline) and post-intervention (within 5-months after baseline measures).
  Hamstring and quadriceps strength will be measured using a handheld dynamometer. Each strength measure will be taken 3 times with the average calculated.
Agility assessment | Agility will be measured at two separate timepoints: pre-intervention (baseline) and post-intervention (within 5-months after baseline measures).
  The Pro-Agility Test utilizes three cones. The farthest cone is sprinted to, the ground is touched with one hand and direction changed back to the starting cone (9.1m sprint). The ground is touched at the starting cone, direction is changed to the 'middle cone' into a 4.6m sprint. Passing the 'middle cone' is the finish line for the test. Each strength measure will be taken 3 times with the average calculated.
Hop testing assessment | Hop performance will be measured at two separate timepoints: pre-intervention (baseline) and post-intervention (within 5-months after baseline measures).
  Participants will complete a single leg hop, triple hop and a timed 6 meter hop
Kinetic jump testing assessment | Kinetic jump performance will be measured at two separate timepoints: pre-intervention (baseline) and post-intervention (within 5-months after baseline measures).
  A countermovement jump and a single leg vertical jump on a force plate platform system.

SECONDARY OUTCOMES:
Injury rates | Duration of spring soccer season, January - May (5 months).
  Injury information provided by coaches and/or parents throughout the spring soccer season.

CONTACTS AND LOCATIONS:
Overall Officials: Shari Liberman, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No